CLINICAL TRIAL: NCT06384131
Title: A Randomized, Blinded, Placebo-Controlled Dose-Ranging Phase 1b Study of the Safety, Pharmacokinetics, and Antiviral Activity of ABI-4334 in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Antiviral Activity of ABI-4334 in Subjects With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-4334-102; 2024-511051-18 (EudraCT Number)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Chronic Hepatitis B
Keywords: cHBV; HBV; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABI-4334 (Active Comparator)
  Interventions: Drug: ABI-4334
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABI-4334 — 10 mg or 50 mg tablets for oral administration
  Arms: ABI-4334
Drug: Placebo — 10 mg or 50 mg tablets for oral administration
  Arms: Placebo

SUMMARY:
This is a randomized, blinded, placebo-controlled, dose-ranging Phase 1b study of the safety, PK, and antiviral activity of ABI-4334 in treatment-naïve or off-treatment chronic Hepatitis B virus (cHBV) subjects that are Hepatitis B e antigen (HBeAg) positive or negative. The study will enroll up to 5 sequential cohorts of 10 subjects each, for a total of up to 50 subjects, randomized 8:2 to receive ABI-4334 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 18.0 and < 35.0 kg/m(2), where BMI = weight (kg)/(height [m])(2) with a minimum body weight of 45 kg
2. Chronic hepatitis B infection, defined as HBV infection for ≥ 6 months documented
3. Treatment-naïve or off-antiviral therapy for ≥ 24 weeks prior to Screening
4. Lack of bridging fibrosis or cirrhosis

Exclusion Criteria:

1. Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis D virus (HDV), acute hepatitis A virus (HAV), or acute hepatitis E virus (HEV)
2. History of liver transplant or evidence of advanced liver disease, cirrhosis, or hepatic decompensation
3. Clinically significant diseases or conditions
4. History of hepatocellular carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ABI-4334 in subjects with cHBV following 28-day multiple oral doses | Through end of study, up to 56 days
  Proportion of subjects with adverse events (AEs), premature treatment discontinuation due to AEs, and abnormal laboratory results

SECONDARY OUTCOMES:
To characterize the PK of ABI-4334 in plasma following 28-day multiple doses in subjects with cHBV | Through treatment period, up to 28 days
  Noncompartmental plasma PK parameters
Changes in HBV DNA in subjects with cHBV following 28-day multiple doses of ABI-4334 | Through treatment period, up to 28 days
  Mean change in log10 HBV DNA between Baseline and Day 28
To characterize the PK of ABI-4334 in plasma following 28-day multiple doses in subjects with cHBV | Through treatment period, up to 28 days
  Area Under Plasma Concentration-Time Curve (AUC) of ABI-4334 in subjects with cHBV
To characterize the PK of ABI-4334 in plasma following 28-day multiple doses in subjects with cHBV | Through treatment period, up to 28 days
  Time to Maximum Plasma Concentration (Tmax) of ABI-4334 in subjects with cHBV
Elimination half-life (t1/2) of ABI-4334 in subjects with cHBV | Through treatment period, up to 28 days
Changes in HBV pregenomic ribonucleic acid (pgRNA) and additional markers of antiviral activity in subjects with cHBV | Through treatment period, up to 28 days
  To evaluate the changes in HBV DNA (IU/mL or Log IU/mL) in subjects with cHBV
Changes in HBV DNA in subjects with cHBV following 28-day multiple doses of ABI-4334 | Through treatment period, up to 28 days
  Proportion of subjects with HBV DNA < lower limit of quantification (LLOQ) and/or limit of detection (LOD)
Changes in HBV DNA in subjects with cHBV following 28-day multiple doses of ABI-4334 | Through treatment period, up to 28 days
  Mean time elapsed to subjects achieving HBV DNA < LLOQ and/or LOD

CONTACTS AND LOCATIONS:
Locations (2):
- ARENSIA Exploratory Medicine Chisinau, Chisinau, Moldova
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No